CLINICAL TRIAL: NCT02755636
Title: Integrative Platform for Primary Care Delivery of Evidence-Based Cancer Risk Behavior Interventions
Brief Title: Pro-Change Population Health Solution
Acronym: PCPHS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pro-Change Behavior Systems (Other)
Collaborators: Community Health Center, Inc. (Industry)
Responsible Party: Principal Investigator, Deborah Levesque, Chief Science Officer, Pro-Change Behavior Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHSN261201500015C
Record Dates: First submitted 2016-03-30; First posted 2016-04-29 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Risk Behavior
Keywords: Health Behavior Change; Primary Health Care; Patient Participation; Provider-Patient Communication; Cluster-Randomized Trial; Mobile Health
MeSH Terms: conditions — Risk-Taking; Patient Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCPHC intervention (Experimental): PCPHC intervention during 6-month intervention period plus study assessments at baseline, 6, and 12 months
  Interventions: Behavioral: PCPHC; Other: Usual care
- Usual care (Active Comparator): Usual primary care plus study assessments at baseline, 6, and 12 months
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: PCPHC — Mobile-delivered health risk intervention (HRI), computer-tailored interventions (CTIs), text messages; provider-delivered one-on-one session guided by clinical dashboard
  Arms: PCPHC intervention
Other: Usual care — Primary care as usual

SUMMARY:
Patients with co-occurring health risk behaviors suffer greater morbidity, disability, and premature death. The Pro-Change Population Health Solution (PCPHS) is a suite of mobile tools designed to assist patients and primary care providers (PCPs) in applying evidence-based principles of health behavior change to reduce four cancer risk behaviors-cigarette smoking, risky drinking, noncompliance with national guidelines for physical activity, and overweight and obesity-and depression among at-risk patients. The intervention is based on the Transtheoretical Model of Behavior Change (TTM, the "stage model") and includes computer-tailored interventions and text messages for patients and a clinical dashboard for providers. The efficacy of the intervention will be assessed in a cluster-randomized trial involving 780 patients recruited from 12 federally qualified health centers randomly assigned to intervention or usual care.

DETAILED DESCRIPTION:
A cluster-randomized design will be used to assess the efficacy of the PCPHS intervention for multiple behavior change for cancer prevention by comparing 6- and 12-month outcomes among 780 primary care patients recruited by 12 federally qualified health clinics randomly assigned to intervention or usual care. A Multiattribute Utility Measurement Approach will be used to ensure that clinics assigned to the two conditions are approximately equivalent on clinic size, patient demographics, and cancer risk behaviors (e.g., rates of smoking, overweight, and obesity). The most similar clinics will be paired, and one clinic within each pair will be assigned to intervention, and the other to usual care.

Patients with an upcoming appointment and who meet study inclusion criteria will be invited to participate in the study, which will begin with an online baseline survey. In addition, patients in the intervention group will complete an online health risk intervention (HRI) that assesses and intervenes on the four cancer risk behaviors targeted in the intervention-cigarette smoking, risky drinking, noncompliance with national guidelines for physical activity, and overweight and obesity-as well depression. It will also assess whether participants have received cancer screenings recommended by age and gender.

After the HRI session, intervention participants will have access to the TTM CTIs targeting their risk factors during the next six months. Patients assigned to the usual care condition will receive care as usual.

Providers at the six clinics assigned to intervention will receive training on the TTM and the clinical dashboard. They will have access to the dashboard via the patient electronic medical record (EMR) during the intervention period, and will be expected to use the dashboard to deliver the one-on-one component of the TTM intervention. The clinical dashboard will:

1. Report whether the participant has received recommended cancer screenings;
2. Summarize data on targeted behavioral risks for cancer;
3. Summarize data on level of depression;
4. For each cancer risk behavior, show stage of change for meeting recommended guidelines; if at least mild depression show stage of change for using healthy strategies to manage depression; and
5. For each cancer risk behavior and depression management, provide stage-matched scripts providers can use to help participants progress to the next stage of change or to prevent relapse to an earlier stage.

Intervention group providers will deliver the dashboard-guided session at the patient's next clinic visit. The dashboard will be updated as the participant completes CTI sessions post-visit. Study participants who return to the clinic for any reason during the intervention period will be flagged, and the provider will use the dashboard to review progress and deliver updated stage-matched guidance.

All study participants will receive an online survey to assess outcomes at 6 and 12 months follow-up. Participants who don't complete the online survey within two weeks will be contacted by a survey research company to complete the survey by phone.

ELIGIBILITY:
Inclusion Criteria:

Has at least one of the following behavioral risk factors for cancer:

1. Cigarette smoker
2. Exceeds recommended limits for alcohol intake
3. Does not meet national guidelines for physical activity
4. Overweight or obese

Exclusion Criteria:

1. Currently pregnant
2. Currently undergoing cancer treatment
3. Serious medical condition that could prevent participation in the study for a full year
4. History of mania, schizophrenia, or other psychoses
5. Admitted to an inpatient mental health facility within the previous 2 years
6. Currently enrolled in the In It to Quit Study at the Community Health Center, Inc.
7. Unable to read English or Spanish
8. Unable to receive text messages

Note: Risky drinkers who screen positive for alcohol dependence will not be eligible for the intervention's risky drinking program, which focuses on limiting drinking to national guidelines. Treatment and control participants who screen positive for alcohol dependence and who are not engaging in any of the other targeted cancer risk behaviors will screen out of the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in number of cancer risk behaviors | Baseline, 12 months
  Change in number of cancer risk behaviors will be computed by taking the difference in the count of the four cancer risk behaviors (cigarette smoking, risky drinking, noncompliance with national guidelines for physical activity, and overweight and obesity) from baseline to 12 months follow-up. At each time point, the index will range from 0 to 4, with each risk behavior scored a "1" if present, and "0" if not present (Prochaska, Prochaska, & Prochaska, 2014).

SECONDARY OUTCOMES:
Change in consumer engagement | Baseline, 12 months
  Change in consumer engagement will be computed by taking the difference in scores on the Altarum Consumer Engagement Measure (Duke, Lynch, Smith, & Winstanley, 2015) from baseline to 12 months follow-up. The measure assesses four dimensions of engagement in healthcare: 1) commitment, 2) informed choice, 3) navigation, and 4) ownership.
Adherence with cancer screenings | 12 months
  Adherence with cancer screenings be the percentage of age- and gender-based U.S. Preventive Services Task Force-recommended screenings received during follow-up.
Change in satisfaction with medical care | Baseline, 12 months
  Change in patient satisfaction will be computed by taking the difference in participant scores on a 1-item global rating of satisfaction with care scale from baseline to 12 months follow-up. The scale is taken from the Consumer Assessment of Healthcare Providers and Systems (CAHPS) survey (Agency for Healthcare Policy and Research, 1999; Hargraves, Hays, & Cleary, 2003).
Change in well-being | Baseline, 12 months
  Change in well-being will be computed by taking the difference in the Cantril Self-Anchoring Scale (Cantril, 1965) from baseline to 12 months follow-up. The measure asks participants to imagine a ladder with steps numbered from zero to ten, with the top representing the best possible life and the bottom representing the worst possible life, and to indicate where they feel their life falls currently and where it will be in five years.
Change in health-related quality of life | Baseline, 12 months
  Change in well-being will be computed by taking the difference in the Centers for Disease Control and Prevention Healthy Days (2000) Core Measures from baseline to 12 months follow-up. The measures assess overall self-rated health, recent physical symptoms, recent mental and emotional distress, and recent activity limitations.

OTHER OUTCOMES:
Change in number of cigarettes smoked per day | Baseline, 12 months
  Will only be assessed among patients smoking at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for smoking cessation | 12 months
  Will only be assessed among patients smoking at baseline (exploratory analysis; study is not powered to find significance)
Change in number of alcoholic drinks per week | Baseline, 12 months
  Will only be assessed among patients exceeding recommended limits at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for drinking within recommended limits | 12 months
  Will only be assessed among patients exceeding recommended limits at baseline (exploratory analysis; study is not powered to find significance)
Change in level of leisure-time exercise | Baseline, 12 months
  Will be assessed using Godin's Leisure-Time Exercise Questionnaire (Godin & Shephard, 1985) only among patients not meeting national guidelines for physical activity at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for meeting national guidelines for physical activity | 6 months, 12 months
  Will only be assessed among patients not meeting national guidelines for physical activity at baseline (exploratory analysis; study is not powered to find significance)
Change in body mass index (BMI) | Baseline, 12 months
  Will be calculated using height and weight only among patients who are overweight (BMI of 25 kg/m2 or higher) at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for engaging in four key behaviors for healthy weight management | 6 months, 12 months
  Progress to the Action stage for 1) reducing daily calorie intake by 500 calories/day, 2) limiting saturated and trans fat intake, 3) managing emotional distress, and 4) meeting national guidelines for physical activity will only be assessed among patients who are overweight (BMI of 25 kg/m2 or higher) at baseline (exploratory analysis; study is not powered to find significance)
Change in level of depression | Baseline, 12 months
  Will be assessed using the Patient Health Questionnaire (PHQ-8) (Kroenke, Strine, Spritzer, Williams, Berry, & Mokdad, 2009) only among patients with at least mild depression (PHQ-8 score of 5 or higher) at baseline (exploratory analysis; study is not powered to find significance)
Progress to the Action stage for managing depression | 6 months, 12 months
  Will only be assessed among patients with at least mild depression (PHQ-8 score of 5 or higher) at baseline (exploratory analysis; study is not powered to find significance)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Levesque, Ph.D., Principal Investigator — Pro-Change Behavior Systems
Locations (2):
- United States (2):
  - Connecticut Health Center, Inc., Middletown, Connecticut
  - Pro-Change Behavior Systems, Inc., South Kingstown, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agency for Healthcare Policy and Research. CAHPS 2.0 survey and reporting kit. Rockville, MD: Agency for Healthcare Policy and Research; 1999.
- [Background] Cantril H. The pattern of human concerns. New Brunswick, NJ: Rutgers University Press; 1965.
- [Background] Centers for Disease Control and Prevention. Measuring Healthy Days: Population Assessment of Health-Related Quality of Life. Atlanta, GA; 2000.
- [Background] Duke CC, Lynch WD, Smith B, Winstanley J. Validity of a New Patient Engagement Measure: The Altarum Consumer Engagement (ACE) Measure. Patient. 2015 Dec;8(6):559-68. doi: 10.1007/s40271-015-0131-2. PMID 26097010
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Graham JW, Flay BR, Johnson CA, Hansen WB, Collins LM. Group comparability: A multiattribute utility measurement approach to the use of random assignment with small numbers of aggregated units. Evaluation Review 1984;8(2):247-60.
- [Background] Hargraves JL, Hays RD, Cleary PD. Psychometric properties of the Consumer Assessment of Health Plans Study (CAHPS) 2.0 adult core survey. Health Serv Res. 2003 Dec;38(6 Pt 1):1509-27. doi: 10.1111/j.1475-6773.2003.00190.x. PMID 14727785
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Prochaska JO, Redding C, Evers K. The Transtheoretical model and stages of change. In: Glanz K, Rimer BK, Viswanath K, editors. Health Behavior and Health Education: Theory, Research and Practice. 4 ed. San Francisco, CA: Jossey-Bass; 2008. p. 97-122.
- [Background] Prochaska J, Prochaska J, Prochaska J. Building a science for multiple-risk behavior change. In: Riekert KA, Ockene JK, Pbert L, editors. The handbook of health behavior change. 4 ed. New York: Springer; 2014. p. 245-67.